CLINICAL TRIAL: NCT02555254
Title: Impact of Speed Of Rewarming After CaRdiac Arrest and ThErapeutic Hypothermia. A Randomized Controlled Pilot Study
Brief Title: Impact of Speed Of Rewarming After CaRdiac Arrest and ThErapeutic Hypothermia
Acronym: ISOCRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHD 013-15
Record Dates: First submitted 2015-09-14; First posted 2015-09-21 (Estimated); Results first posted 2025-05-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Heart Arrest; Cardiac Arrest; Hypothermia
Keywords: cardiac arrest; targeted temperature management; hypothermia induced; shockable rhythm
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low speed of rewarming (Experimental): Patients will be placed in targeted temperature controlled at 33°C for 24 hours. Then, intervention will be proceeded after randomization: slowly rewarmed (0.25°C/h) to targeted temperature controlled at 37°C for 24 hours.
  Interventions: Procedure: Low Speed of Rewarming
- Fast speed of rewarming (Experimental): Patients will be placed in targeted temperature controlled at 33°C for 24 hours. hen, intervention will be proceeded after randomization: fastly rewarmed (0.50°C/h) for targeted temperature controlled at 37°C for 24 hours.
  Interventions: Procedure: High Speed of Rewarming

INTERVENTIONS:
Procedure: Low Speed of Rewarming — Speed of rewarming will be at 0.25°C/h with specific temperature controlled external device
  Arms: Low speed of rewarming
Procedure: High Speed of Rewarming — Speed of rewarming will be at 0.50°C/h with specific temperature controlled external device
  Arms: Fast speed of rewarming

SUMMARY:
Comparing the production of interleukin 6 (inflammatory cytokine) in two heating speed (slow rewarming rate: 0.25 ° C / h or fast rewarming rate 0.50 ° C / h) at the completion of a period of targeted temperature at 33°C after cardiac arrest supported by shockable rhythm and successfully resuscitated.

DETAILED DESCRIPTION:
Cardiac arrest (CA) is at present a major cause of mortality as well as a cause of disability for the surviving victims. In France, every year counts as 50,000 cardiac arrests responsible for 40 000 deaths. Thus, less than 20% of patients with heart failure discharged home. Then these patients had impaired quality of life associated with symptoms of fatigue, stress, anxiety hindering the resumption of business activity including. The prognosis is related in part to the initial cardiac rhythm present at the establishment of specialized resuscitation.

Recent progress in improving mortality and neurological outcome has been achieved over the last decade with systematic implementation of a period of targeted temperature management between 32 and 34 ° C (TTM 32-34) in patients with cardiac arrest and who benefited from the completion of at least one external electrical shock when help arrived. The mechanisms underlying this improvement of neurological prognosis are many, but mainly related to an attenuation of post resuscitation syndrome that combines in one hand an inflammatory response (mediated by pro-inflammatory cytokines including interleukin 6) and secondly the formation of reperfusion injury related to the production of radical oxygen species (free radicals).

While some studies have shown the feasibility of induction of this TTM 32-34 in prehospital conditions, no prospective study has evaluated the significant speed of warming in the end. An observational study in which the heating was carried passively, found that patients with an extended heating period (600 minutes) had a worse neurological outcome than patients with a duration of shorter warming (479 minutes) while a second retrospective study concluded the opposite in case of active warming . Besides the fact that these studies were observational, in the two originals randomized studies on TTM 32-34 in CA, the rate of warming was not like:

* Objective 6 hours with active warming is 0.5 ° C / h in the Australian study with an OR of 5.25 (1.47 - 18.76) for the neurological prognosis
* Objective 8 hours with passive warming of 0.37 ° C / h in the European study with an OR of 1.4 (1.08 - 1.81) for the neurological prognosis Although populations of two studies are obviously not comparable, it is possible that suboptimal speed of rewarming could mitigate some of the gain related to the implementation of TTM 32-34.

In this context, investigators propose to conduct a randomized, single-center pilot study comparing a fast warming in a slow warming when performing a TTM 33 patients presented with a shockable cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been supported for a shockable cardiac arrest with successful resuscitation.
* Coma persistent at ICU admission (Glasgow score less than or equal to 8) in the absence of sedation. If the patient is sedated in ICU admission, the glasgow score will be held the last evaluated by the doctor who provided the pre-hospital care of the patient score.
* Body temperature> 33 ° C
* Specific device used to targeted temperature management at 33°C

Exclusion Criteria:

* Lack of witness of cardiac arrest.
* Duration of no-flow> 10 minutes (time between the onset of cardiac arrest and the start of external cardiac massage).
* Duration of low-flow> 60 minutes (the period between the start of external cardiac massage and recovery of an effective cardiac activity).
* Major hemodynamic instability (dose norepinephrine and / or epinephrine > 1 µg / kg / min to maintain MAP> 65 mmHg).
* Time between cardiac arrest and more than 480 minutes inclusion
* Moribund.
* Presence of histologically confirmed cirrhosis of Child class C.
* Patient treatment in blocking the production of Il6 (Ro-tocilizumab or Actemra ®)
* Patient under corticosteroid treatment (dose> 5 mg of prednisolone equivalent)
* Pregnant woman, parturient or lactating.
* Inpatient without consent and / or deprived of liberty by a court decision.
* Patient under guardianship
* Inclusion in advance a research protocol with the draw, and whose primary endpoint is on interleukin-6.
* Lack of social security.
* Refusal of the trusted person or patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2020-05-17 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Baptiste Lascarrou, MD, Study Chair — Nantes University Hospital
Locations (1):
- Colin Gwenhael, La Roche-sur-Yon, France

REFERENCES:
- [Background] Pouplet C, Colin G, Guichard E, Reignier J, Le Gouge A, Martin S, Lacherade JC, Lascarrou JB; AfterROSC network. The accuracy of various neuro-prognostication algorithms and the added value of neurofilament light chain dosage for patients resuscitated from shockable cardiac arrest: An ancillary analysis of the ISOCRATE study. Resuscitation. 2022 Feb;171:1-7. doi: 10.1016/j.resuscitation.2021.12.009. Epub 2021 Dec 13. PMID 34915084
- [Result] Lascarrou JB, Guichard E, Reignier J, Le Gouge A, Pouplet C, Martin S, Lacherade JC, Colin G; AfterROSC network. Impact of rewarming rate on interleukin-6 levels in patients with shockable cardiac arrest receiving targeted temperature management at 33 degrees C: the ISOCRATE pilot randomized controlled trial. Crit Care. 2021 Dec 17;25(1):434. doi: 10.1186/s13054-021-03842-9. PMID 34920723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were admitted in medical-surgical ICU at local hospital of La Roche sur Yon, France. and assessed for eligibility between February 12, 2016, and May 15, 2020.
  Patients were included at ICU admission. Randomization occurred at the end of the hypothermia maintenance phase, i.e., 18-24 h after reaching 33 °C.
Pre-assignment Details: Of 160 patients assessed for eligibility, 102 did not meet inclusion criteria, 58 were included and 50 were randomized
Groups:
- Rewarming at 0.5°C/h: Speed of rewarming will be at 0.5°C/h with specific temperature controlled external device
- Rewarming at 0.25°C/h: Speed of rewarming will be at 0.25°C/h with specific temperature controlled external device
Period: Overall Study
Arm/Group | Rewarming at 0.5°C/h | Rewarming at 0.25°C/h
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rewarming at 0.50°C/h: Speed of rewarming will be at 0.50°C/h with specific temperature controlled external device
- Total: Total of all reporting groups
Arm/Group | Rewarming at 0.25°C/h | Rewarming at 0.50°C/h | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.2 [52.2 to 72.4] | 53.8 [48.2 to 70.0] | 61 [48.2 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data not collected in the study Population: Data not collected

OUTCOME MEASURES:

1. Primary Outcome: Changes in Serum Il6 Levels Over the 48 Hours Following Achievement of the Thermal Target
Description: Median AUC for serum IL6 levels over time
Time Frame: 48 hours
Population: One patient died between H32 and H40 and was not included in this analysis given the absence of data for the H40 and H48 time points.
Measure: Median (Inter-Quartile Range); unit: pg/mL*h
Arm/Group | Rewarming at 0.25°C/h | Rewarming at 0.50°C/h
Number analyzed (Participants) | 24 | 25
pg/mL*h | 12389 [7256 to 37200] | 8859 [6825 to 18088]
Statistical Analysis 1: Comparison: Rewarming at 0.25°C/h vs Rewarming at 0.50°C/h; Test type: Superiority; p = 0.55, Wilcoxon's rank test

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Description: Adverse events were not collected
Arm/Group | Rewarming at 0.25°C/h | Rewarming at 0.50°C/h
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT02555254/Prot_SAP_000.pdf